CLINICAL TRIAL: NCT04471025
Title: A Prospective, Randomized, Observer-Blinded Comparison Between Single And Double Operator In Ultrasound Guided Infraclavicular Block: Jedi Grip Versus Conventional Double Operator Technique
Brief Title: Jedi Grip Versus Double Operator Technique For Ultrasound Guided Infraclavicular Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, ismail aytaç, assistant professor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-18-1935
Record Dates: First submitted 2020-07-04; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Ultrasound; Nerve Block
Keywords: Jedi Grip; Ultrasound guided infraclavicular block

STUDY DESIGN:
Intervention Model Description: single-center, prospective, randomized into two goups: Jedi grip versus conventional double operator technique
Who Masked: Outcomes Assessor
Masking Description: After completion of the block, a single blinded observer recorded demographic data and evaluated the block characteristics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): USG guided infraclavicular block with single operator jedi grip technique
  Interventions: Procedure: USG guided infraclavicular block
- Group 2 (Active Comparator): USG guided infraclavicular block with conventional double operator technique
  Interventions: Procedure: USG guided infraclavicular block

INTERVENTIONS:
Procedure: USG guided infraclavicular block — USG guided infraclavicular block was applied to patients either by conventional two-person technique or by one person Jedi technique according to the allocated group. On Group I single operator controlled the probe with one hand while controlling the needle and the syringe on the other hand with the Jedi technique. The needle was held between the index finger and the middle phalanx of the middle finger, and the syringe was held with fingers 4 and 5, with the plunger part to the thumb in the palm. On Group II, operator used the probe and needle with different hands while an assistant controlling the syringe to aspirate or inject local anesthetic.

SUMMARY:
The investigators aimed to compare the block characteristics of the single operator "jedi grip" technique and the conventional double operator technique.

DETAILED DESCRIPTION:
Patients undergoing hand, wrist, elbow and forearm surgery randomly assigned two groups (Group I: Jedi grip and Group II: Conventional double operator technique). By a blind observer, the block characteristics were evaluated and recorded .

ELIGIBILITY:
Inclusion Criteria:

* undergoing elective hand, wrist and forearm surgery

Exclusion Criteria:

* hepatic or renal failure
* serious cardiac or pulmoner disease
* local or systemic infection
* sepsis
* coagulation disorder
* neurological, muscular or psychiatric disease
* body mass index (BMI) below 18.5 or above 35
* drug and substance abuse
* pregnancy
* refusal of regional anesthesia
* history of allergy to local anesthetics
* mental-motor retardation (inability to consent or assess the visual analog scale(VAS) pain score)
* preoperative long-term NSAIDs or opioid use.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
block performance time | during block application
  teh sum of imaging and needling time
block success | during surgery
  incidence of ( %) surgery with successful anesthesia

SECONDARY OUTCOMES:
Sensory block onset time | before surgery
  Sensory blockage was evaluated and graded; from lateral to the forearm, the volar face of the thumb, volar face of the 5th finger and lateral side of the hand back; for musculocutaneous, median, ulnar and radial nerves, respectively. Graduation was according to a previously validated 3-point scale using a cold test: 0 = no block, 1 = analgesia (patient can feel touch, not cold), and 2 = anesthesia (patient cannot feel touch)
motor block onset time | before surgery
  blockage was evaluated and graded; with elbow flexion, thumb abduction, thumb opposition, thumb adduction for musculocutaneous, radial, median, ulnar nerves respectively. Motor blockage graduation was also according to a (validated) 3-point scale: 0 = no block, 1 = paresis and 2 = paralysis.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Aytac, Principal Investigator — Ankara City Hospital Anesthesiology Department
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pappin D, Christie I. The Jedi Grip: a novel technique for administering local anaesthetic in ultrasound-guided regional anaesthesia. Anaesthesia. 2011 Sep;66(9):845. doi: 10.1111/j.1365-2044.2011.06845.x. No abstract available. PMID 21831086